CLINICAL TRIAL: NCT04664647
Title: The Clinical Features of Combined Central and Peripheral Demyelination
Acronym: CCPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, haojunwei, Princple investigation, Xuanwu Hospital, Beijing
Other Study IDs: haojunwei1
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Combined Central and Peripheral Demyelination Disease
Keywords: CCPD; clinical features; antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CCPD: Inclusion criteria：
  1. Criteria for central nervous system involvement: T2 high-signal intensity lesions in the brain, or spinal cord on MRI, or visual-evoked potentials(VEPs) abnormalities.
  2. Criteria for peripheral nervous system involvement: conduction delay, conduction block, temporal dispersion or F-wave abnormalities, suggesting peripheral demyelinating neuropathy regarding nerve conduction studies (NCS). In the present study, it was compulsory for at least two nerves between the median, ulnar, tibial and peroneal nerves to have abnormal findings indicating demyelination.
  Exclusion criterion:
  Secondary demyelinating diseases or changes.

SUMMARY:
The investigators conduct this study to clarify the clinical features and to evaluate the prevalence of anti-nodal/paranodal antibodies of patients with combined central and peripheral demyelination (CCPD) .

DETAILED DESCRIPTION:
The investigators will review the clinical manifestation, laboratory test results, electrophysiological examination and neuroimaging findings of patients with CCPD. And we will detect antibodies to aquaporin 4(AQP4), myelin oligodendrocyte glycoprotein (MOG), neurofascin-155 (Nfasc155), neurofascin-186 (Nfasc186), and myelin-associated glycoprotein (MAG) in patients with CCPD.

ELIGIBILITY:
Inclusion Criteria:

1. T2 high-signal intensity lesions in the brain or spinal cord on MRI, or visual-evoked potentials(VEPs) abnormalities.
2. conduction delay, conduction block, temporal dispersion or F-wave abnormalities, suggesting peripheral demyelinating neuropathy regarding nerve conduction studies (NCS).

Exclusion Criteria:

1. infectious diseases(e.g., human T lymphocyte trophic virus type1-associated myelopathy, syphilis, neuroborreliosis, HIV infection or progressive multifocal leukoencephalopathy)
2. pre-existing inflammatory diseases (e.g., sarcoidosis, Behçet's disease, Sjögren's syndrome, vasculitis or other collagen diseases)
3. mitochondrial disease
4. metabolic/toxic diseases (e.g., vitamin deficiency, amyloidosis, chronic alcoholism, diabetes mellitus or subacute myelo-opticoneuropathy due to clioquinol intoxication
5. cervical spondylotic myelopathy
6. syringomyelia
7. spinocerebellar degeneration
8. multiple myeloma, other tumors
9. inherited diseases (e.g., leucodystrophies)
10. cerebrovascular disease
11. non-specific lesions on T2-weighted MRI (e.g., leucoaraiosis).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have combined central and peripheral demyelination
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Laboratory findings of nodal/paranodal antibodies in blood of patients with CCPD | Day 1 post-gathering information of patients in hospital medical record system
  These antibody including anti-neurofascin 155(NF155) et.al.

SECONDARY OUTCOMES:
Demographic characteristics | Day 1 post-gathering information of patients in hospital medical record system
  The demographic characteristics of patients with CCPD such as age,sex,and et.al
Neurological symptoms and signs | Day 1 post-gathering information of patients in hospital medical record system
  The neurological symptoms and signs of patients with CCPD
Laboratory findings of blood and cerebrospinal fluid | Day 1 post-gathering information of patients in hospital medical record system
  Laboratory findings of blood and cerebrospinal fluid of patients with CCPD such as C reactive protein et.al in blood and protein et.al in cerebrospinal fluid
Neuroimaging and VEPs findings | Day 1 post-gathering information of patients in hospital medical record system
  Neuroimaging and VEPs findings of patients with CCPD
Nerve conduction study findings | Day 1 post-gathering information of patients in hospital medical record system
  Nerve conduction study findings of patients with CCPD

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, Principal Investigator — Xuanwu Hospital, Beijing

REFERENCES:
- [Background] Cortese A, Franciotta D, Alfonsi E, Visigalli N, Zardini E, Diamanti L, Prunetti P, Osera C, Gastaldi M, Berzero G, Pichiecchio A, Piccolo G, Lozza A, Piscosquito G, Salsano E, Ceroni M, Moglia A, Bono G, Pareyson D, Marchioni E. Combined central and peripheral demyelination: Clinical features, diagnostic findings, and treatment. J Neurol Sci. 2016 Apr 15;363:182-7. doi: 10.1016/j.jns.2016.02.022. Epub 2016 Feb 10. PMID 27000248
- [Background] Ogata H, Matsuse D, Yamasaki R, Kawamura N, Matsushita T, Yonekawa T, Hirotani M, Murai H, Kira J. A nationwide survey of combined central and peripheral demyelination in Japan. J Neurol Neurosurg Psychiatry. 2016 Jan;87(1):29-36. doi: 10.1136/jnnp-2014-309831. Epub 2015 Feb 11. PMID 25673872
- [Background] Wang YQ, Chen H, Zhuang WP, Li HL. The clinical features of combined central and peripheral demyelination in Chinese patients. J Neuroimmunol. 2018 Apr 15;317:32-36. doi: 10.1016/j.jneuroim.2018.02.006. Epub 2018 Feb 9. PMID 29501083
- [Background] Nave KA, Werner HB. Myelination of the nervous system: mechanisms and functions. Annu Rev Cell Dev Biol. 2014;30:503-33. doi: 10.1146/annurev-cellbio-100913-013101. PMID 25288117
- [Background] Stathopoulos P, Alexopoulos H, Dalakas MC. Autoimmune antigenic targets at the node of Ranvier in demyelinating disorders. Nat Rev Neurol. 2015 Mar;11(3):143-56. doi: 10.1038/nrneurol.2014.260. Epub 2015 Jan 27. PMID 25623793